CLINICAL TRIAL: NCT00003899
Title: High-Dose Consolidation With Escalating Doses of Melphalan and Thiotepa for Stage IV Breast Cancer
Brief Title: Chemotherapy Plus Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1343.00; FHCRC-1343.00; NCI-H99-0032; CDR000006707 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2010-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Filgrastim; Cyclophosphamide; Melphalan; Paclitaxel; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: melphalan
Drug: paclitaxel
Drug: thiotepa
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow or peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of melphalan and thiotepa plus bone marrow or peripheral stem cell transplantation in treating patients who have recurrent or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of melphalan and thiopeta in patients with recurrent or refractory solid tumors. II. Evaluate the overall survival and response rate in these patients.

OUTLINE: This is a dose escalation study. Patients receive cyclophosphamide IV over 1 hour on day 1 and paclitaxel IV over 4 or 24 hours on day 2, followed by daily filgrastim (G-CSF) subcutaneously beginning on day 3 and continuing through day 7 or until WBCs are greater than 100,000 cells/mm3. Peripheral blood stem cells (PBSC) or autologous bone marrow is collected on days 5-7. At 30-50 days following mobilization, patients receive melphalan IV over 15-60 minutes on days -5 and -4 and thiotepa IV over 2 hours on days -3 and -2, followed by autologous bone marrow transplantation or PBSC infusion on day 0. Sequential dose escalation of melphalan is followed by sequential dose escalation of thiotepa. Dose escalation in cohorts of 5 patients each continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 4, 3 of 7, 4 of 11, or 5 of 15 patients experience dose limiting toxicity. Patients are followed at 60 days and at 12 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed solid tumor Metastatic disease Recurrent or refractory Pleural effusions allowed, if controlled Brain metastases allowed, if symptoms controlled and negative MRI

PATIENT CHARACTERISTICS: Age: 18 to 65 Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 No uncontrolled bleeding Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT and/or SGPT less than 3 times normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: Normal EKG Ejection fraction at least 45% Patients with abnormal EKG, history of myocardial infarction, unstable angina, congestive heart failure, or prior cumulative anthracycline dose of at least 250 mg/m2, must have a left ventricular ejection fraction performed No congestive heart failure or uncontrolled hypertension Pulmonary: DLCO greater than 60% No pneumonia No asthma, even if controlled Neurologic: No dementia or altered mental status Other: No active infection (e.g., peritonitis, wound abscess) HIV negative No prior cyclophosphamide induced hemorrhagic cystitis No serious concurrent systemic disease (e.g., diabetes mellitus, hypothyroidism) No other active malignancies Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No other concurrent chemotherapy Endocrine therapy: Concurrent hormonal therapy allowed Radiotherapy: No concurrent radiotherapy Surgery: At least 2 weeks since prior surgery and recovered

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01; Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States